CLINICAL TRIAL: NCT04391166
Title: Validity of at Home Visual Acuity Measurements for Telemedicine During Corona Virus (COVID-19) Pandemic
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sapna Gangaputra, Assistant Professor of Ophthalmology, Vanderbilt University Medical Center
Other Study IDs: 200826
Record Dates: First submitted 2020-05-15; First posted 2020-05-18 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Visual Impairment
Keywords: ETDRS Visual acuity
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non invasive visual acuity testing — This will be visual acuity at home and visual acuity in clinic both using an ETDRS chart.

SUMMARY:
Prompted by the current COVID-19 pandemic, the American Academy of Ophthalmology has recommended the use of telemedicine to continue ophthalmic care while maintaining patient and provider social distancing. As part of remote examinations, patients may be expected to perform home eye testing for visual acuity and the use of various home visual acuity charts have been proposed to provide clinicians with this vital data. However, the use of home visual acuity exams has not been validated in our patient population. This project aims to determine the efficacy and validity of measuring visual acuity at home with a printed-out ETDRS chart.

DETAILED DESCRIPTION:
Project Title Validity of Home Visual Acuity Measurements with an ETDRS Chart

Project Summary Prompted by the current COVID-19 pandemic, the American Academy of Ophthalmology has recommended the use of telemedicine to continue ophthalmic care while maintaining patient and provider social distancing. As part of remote examinations, patients may be expected to perform home eye testing for visual acuity and the use of various home visual acuity charts have been proposed to provide clinicians with this vital data. However, the use of home visual acuity exams has not been validated in our patient population. This project aims to determine the efficacy and validity of measuring visual acuity at home with a printed-out ETDRS chart.

Project Description Rationale: Many ophthalmology visits are being conducted remotely via telehealth. The use of home ETDRS charts is being proposed for patients to report their visual acuity. However, the efficacy and validity of this method in our population should be determined.

Objective: Determine the efficacy and validity of measuring visual acuity at home with a printed-out ETDRS chart in the population served by Vanderbilt Eye Institute. Our hypothesis is that measuring visual acuity at home with a printed-out ETDRS is non-inferior to visual acuity measurements by a trained technician in the clinic.

Methodology: The study population will include patients scheduled for in-person visits for various subspecialties (Glaucoma, Retina/Uveitis, Pediatrics and Cornea) at Vanderbilt Eye Institute's (VEI) Nashville campus during the period of 4/27/20-5/27/20. Patients will be excluded if they have a last best corrected visual acuity worse than 20/200, have not activated a My Health at Vanderbilt (MHAV) account, or do not speak English. Patients will also need to be between the ages of 18-90 to Approximately one week prior to their appointments, patients will be called to obtain e-consent and provide detailed instructions for measuring best corrected visual acuity at home with the ETDRS chart that is calibrated for 5 feet. Instructions will also be sent via MHAV along with the ETDRS chart and the consent form. Data collected will include age, sex, and primary ophthalmological diagnosis as well as last measured Snellen visual acuity (+/-3months). The department, provider, and date of the in-person appointment will also be collected. Patients will be instructed to complete a home visual acuity check two-four days prior to appointment and send a message through MHAV with the results. Participants will record the smallest full line ( 5 letters) in each eye that they can read. If a message is not received two days prior to the appointment, a research assistant will call the patient back to reconfirm the plan. At the in-person visit, patients will begin their encounter with an ETDRS assessment at VEI, using the ETDRS chart at 20 feet. Again, the full line of 5 letters read will be used for analysis. Patients will receive a survey to be completed in clinic with a 5-point Likert scale to rate the ease of home visual acuity as well as a short response question about barriers to assessment.

Data Management and Analysis: Data will be collected from the electronic health record (EHR) and kept in a password-protected deidentified Excel document. Visual acuities will be converted to logMAR for analysis.

Ethical Considerations: There are no ethical considerations to report.

Barriers to Home Visual acuity testing

* Poor/no access to the technical requirements - computer, printer, internet
* Do not feel confident of being able to test vision accurately at home
* Attempted to test vision at home but was unable to follow instructions completely
* Do not want to try it at home, medical procedures should be done in a clinic
* Vision too poor to perform these tasks

The Home visual acuity test was easy to set up and perform

1. Strongly disagree
2. Disagree
3. Neither agree nor disagree
4. Agree
5. Strongly agree

ELIGIBILITY:
Inclusion Criteria:

* The study population will include patients scheduled for in-person visits for various subspecialties (Glaucoma, Retina/Uveitis, pediatrics and Cornea) at Vanderbilt Eye Institute's (VEI) Nashville campus during the period of 4/27/20-5/8/20.

Exclusion Criteria:

* Patients will be excluded if they have a last best corrected visual acuity worse than 20/200.
* If they have not activated a My Health at Vanderbilt (MHAV) account
* If they do not speak English.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include patients scheduled for in-person visits for various subspecialties (Glaucoma, Retina/Uveitis, pediatrics and Cornea) at Vanderbilt Eye Institute's (VEI) Nashville campus during the period of 4/27/20-5/8/20.
  Between the ages of 18-90.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) Per Eye | From the time they sign the consent until we take their BCVA in clinic. Approximately 1-2 weeks.
  Best Visual Acuity per eye

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt Eye Institute, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No